CLINICAL TRIAL: NCT05655741
Title: Developing Best Practice for Genomic Bereavement Care in Pregnancy Loss: A Modified Delphi Consensus Study.
Brief Title: Modified Delphi for Genomic Bereavement Care
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Genomic Medicine Services Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: CG22/151813
Record Dates: First submitted 2022-09-28; First posted 2022-12-19 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Fetal Anomaly; Bereavement; Genetic Disease
MeSH Terms: conditions — Congenital Abnormalities; Genetic Diseases, Inborn | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi Panel: Participants who meet the inclusion criteria ,who are willing to complete the 3 questionnaires within the study.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will be asked to complete a series of 3 questionnaires that will be used to gain insight into the current expert consensus for Genomic Bereavement care for Pregnancy Loss.
  The 2nd and 3rd Questionnaire will be modified from the first to try to generate consensus, depending on the answers from the previous round.

SUMMARY:
It is estimated that 1 in 4 pregnancies end in loss, be these early miscarriages, ectopic pregnancies, or later intrauterine losses for any reason. Genomics is a major part of pregnancy loss, and clinicians want to offer the best and most appropriate test available to women and their families, whilst ensuring that there is equity in the access to this testing, so that no family goes through a loss without the right support and information. Whilst there is limited information to inform professionals as to how to incorporate genomics into bereavement care there is a need to identify current expert consensus as to how this should be performed, in order to make recommendations for best practice.

DETAILED DESCRIPTION:
There is a lack of guidance available as to how to care for women and families who suffer a pregnancy loss where fetal anomalies have been found and a genetic cause is suspected. As it is estimated that 1 in 4 pregnancies end in loss, these families make up a significant proportion of the population that maternity services care for and with no consensus in this area many families may have a poor experience.

As the field of genomics rapidly advances, it is important that patient care reflects the changes in practice and that the most appropriate tests and support are offered. All aspects of patient care will be reviewed including diagnosis, delivery, laboratory investigations, postnatal care and follow up in future pregnancies. The role of the genomics midwife will be explored and the role of the bereavement midwife will be further defined when it comes to support following pregnancy loss where there is likely an underlying genomic cause.

The aim of this modified delphi study is to understand what the current expert consensus is for genomic bereavement care. Using this, best practice guidance will be written that can be used within the NHS to better support families who suffer pregnancy loss during this pregnancy and in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participants must belong to one of the relevant stakeholder groups; Maternal and fetal medicine consultants or obstetricians with a special interest in fetal medicine, Clinical geneticists with an interest in prenatal genomics, Perinatal pathologists Clinical scientists with an interest in genomics, Bereavement midwives.

Exclusion Criteria:

* Nil if inclusion criteria are met

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be contacted via email with an advert for the study in order to declare an expression of interest. Relevant groups will include; BMFMS members, Fetal Genomics Group steering group for those with prenatal interests, BRIPPA members for pathologists with an interest in perinatal pathology, Laboratory leads for each GMSA, a bereavement midwife from each GMSA.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Identify consensus for best practice for genomic bereavement care | 26 weeks
  Consensus will be achieved if >80% of participants agree or strongly agree with the statement using a 5 point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Hyland, MBBS, Principal Investigator — Leeds Teaching Hospitals Trust
Locations (1):
- Leeds Teaching Hospitals Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No